CLINICAL TRIAL: NCT04204811
Title: A Pilot Project to Evaluate Feasibility and Patient Experience of Prehabilitation Care for Women With Advanced Ovarian Cancer Undergoing Neoadjuvant Chemotherapy
Brief Title: Prehabilitation Care for Women With Advanced Ovarian Cancer Receiving Neoadjuvant Chemotherapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-347
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer; Stage III Ovarian Cancer; Stage IV Ovarian Cancer; Primary Peritoneal Carcinoma; Fallopian Tube Carcinoma; Fallopian Tube Cancer
Keywords: Ovarian Cancer; Primary peritoneal carcinoma; Fallopian tube cancer; 19-347; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with Ovarian Cancer (Experimental): Participants are diagnosed with Stage III or Stage IV ovarian carcinoma (which includes primary peritoneal carcinoma or fallopian tube carcinoma)
  Interventions: Other: Prehabilitation

INTERVENTIONS:
Other: Prehabilitation — A program of personalized independent home exercises are outline for participants to complete daily. Prehabilitation coaching will continue weekly until admission for surgical tumor debulking or termination of neoadjuvant treatment for any reason.

SUMMARY:
The purpose of this study is evaluate whether a prehabilitation program is feasible and useful for women with advanced ovarian cancer receiving chemotherapy in preparation for debulking surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be diagnosed with Stage III or Stage IV ovarian carcinoma (which includes primary peritoneal carcinoma or fallopian rube carcinoma)
* All subjects must be enrolled within 90 days of diagnosis
* No prior treatment for ovarian carcinoma
* All subjects have agreed to a treatment plan of neoadjuvant chemotherapy and subsequent planned interval debulking surgery with an MSKCC surgeon
* Participants must be initiating treatment at Gynecologic Medical Oncology clinics at MSKCC Manhattan
* Proficiency in English in the determination of the investigators of by patient self-report

Exclusion Criteria:

* Patient under age 18
* Prior treatment for ovarian cancer
* Second opinion visit only
* Immediate surgery plan without neoadjuvant treatment
* No intended surgical plan
* Chemotherapy administration exclusively planned at MSKCC regional site
* Patient unwilling to sign consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2026-12-16 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Median completion of participants | Up to 1 year
  Study will be considered feasible if the cohort has a median completion of 70% or more

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Gillis, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org